CLINICAL TRIAL: NCT05270369
Title: Effects of Group-based and Digitally Delivered Cognitive Behavioural Therapy for Insomnia (CBT-I) in Youth: a Randomised Controlled Trial
Brief Title: Effects of Group-based and Digitally Delivered CBT-I in Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other); University of Oxford (Other)
Responsible Party: Principal Investigator, Dr. Shirley Xin Li, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA200037
Record Dates: First submitted 2022-02-14; First posted 2022-03-08 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Insomnia
Keywords: youth; sleep; insomnia; CBT-I
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- digital cognitive behavioural therapy for insomnia (CBTI) (Experimental): The digital CBTI group will receive 6-session on their smartphone application
  Interventions: Behavioral: digital CBTI
- group cognitive behavioural therapy for insomnia (CBTI) (Experimental): The group CBTI will receive 6-session CBTI in group
  Interventions: Behavioral: group CBTI
- waitlist (No Intervention): The waitlist group will receive treatment sessions after about 10 weeks' time

INTERVENTIONS:
Behavioral: digital CBTI — The app-based intervention will consists of 6 weekly sessions and will be delivered within a 10-week window. The treatment components aim to address the behavioural, cognitive and physiological factors perpetuating insomnia whilst considering the sleep and circadian features in adolescents and developmental context with the following key elements: psycho-education about sleep, circadian rhythm and sleep hygiene, stimulus control, sleep restriction, relaxation training, structured worry time, cognitive restructuring (targeting sleep-related dysfunctional cognitions), and relapse prevention
  Arms: digital cognitive behavioural therapy for insomnia (CBTI)
Behavioral: group CBTI — The group-based CBT-I intervention will consist of 6 weekly sessions (90-min, 5-8 adolescents in each group) and will be delivered within a 10-week window. The treatment components aim to address the behavioural, cognitive and physiological factors perpetuating insomnia whilst considering the sleep and circadian features in adolescents and developmental context with the following key elements: psycho-education about sleep, circadian rhythm and sleep hygiene, stimulus control, sleep restriction, relaxation training, structured worry time, cognitive restructuring (targeting sleep-related dysfunctional cognitions), and relapse prevention
  Arms: group cognitive behavioural therapy for insomnia (CBTI)

SUMMARY:
Adolescence is a critical transitional stage characterised by a cascade of developmental changes in biological, cognitive, and psychological functioning. Sleep problems, particularly insomnia, are prevalent in adolescents, with a prevalence rate as high as 36%. Insomnia symptoms, presented as the problems initiating sleep or maintaining sleep, have often been reported in association with adverse outcomes in adolescents, including an increased risk of developing depression, anxiety, interpersonal problems, somatic health problems, self-harm and suicidal ideation. This study tests the efficacy of cognitive behavioural therapy for insomnia (CBT-I) in reducing insomnia severity in youth with insomnia.

ELIGIBILITY:
Inclusion Criteria:

* (1) Chinese aged 12-20 years old (an age range that was similarly adopted in the previous studies to cover a wider developmental span in adolescence);
* (2) Written informed consent of participation into the study is given by the participant and his/her parent or guardian (for those aged under 18);
* (3) Willing to comply with the study protocol;
* (4) Meeting the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnostic criteria of insomnia disorder and with a score on Insomnia Severity Index (ISI) - 9 (suggested cut-off for adolescents)

Exclusion Criteria:

* (1) A current diagnosis of substance abuse or dependence; a current or past history of manic or hypomanic episode, schizophrenia spectrum disorders, neurodevelopmental disorders, organic mental disorders, or intellectual disabilities;
* (2) Having a prominent medical condition known to interfere with sleep continuity and quality (e.g. eczema, gastro-oesophageal reflux disease);
* (3) Having a clinically diagnosed sleep disorder that may potentially contribute to a disruption in sleep continuity and quality, such as narcolepsy, sleep-disordered breathing, and restless leg syndrome, as ascertained by the Structured Interview for Sleep Patterns and Disorders (DISP), a validated structured diagnostic interview to assess major sleep disorders according to the International Classification of Sleep Disorder (ICSD) criteria;
* (4) Concurrent, regular use of medications(s) known to affect sleep continuity and quality including both western medications (e.g. hypnotics, steroids) and over-the-counter (OTC) medications (e.g. melatonin, Traditional Chinese Medicine, TCM);
* (5) Having been enrolled in any other clinical trial investigational products within one month at the entry of the study;
* (6) In the opinion of the research clinician, having a clinically significant suicidality (presence of suicidal ideation with a plan or an attempt) as assessed by Mini-International Neuropsychiatric Interview (MINI);
* (7) Currently receiving any structured psychotherapy;
* (8) With hearing or speech deficit; (9) Night shift worker.

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 159 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Change of insomnia symptoms | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Insomnia symptoms measured by Insomnia Severity Index (ISI). ISI is a 7-item self-rated scale. Possible scores range from 0 to 28, with higher scores indicating higher insomnia severity.

SECONDARY OUTCOMES:
Change in Sleep Quality | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Pittsburgh Sleep Quality Index (PSQI) is a self-rated scale consisting of 19 questions. All items are combined to form seven component scores on different aspects of sleep quality, each of which ranges from 0 to 3 points with higher scores representing more sleep disturbance. The seven component scores are added to one global score, which ranges from 0 to 21, with higher scores indicating more difficulties with sleep.
Change of Sleep Diary Measure - Time in Bed (TIB) | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: time in bed (TIB) in hours
Change of Sleep Diary Measure - Total Sleep Time (TST) | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: total sleep time (TST) in hours
Change of Sleep Diary Measure - Sleep Onset Latency (SOL) | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: sleep onset latency (SOL) in mins
Change of Sleep Diary Measure - Wake After Sleep Onset (WASO) | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: wake after sleep onset (WASO) in mins
Change of Sleep Diary Measure - Sleep Efficiency (SE) | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: sleep efficiency (SE), which is calculated by total sleep time divided by total time in bed, %
Change in Objective Sleep Measures - Time in Bed (TIB) | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: time in bed (TIB) in hours
Change in Objective Sleep Measures - Total Sleep Time (TST) | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: total sleep time (TST) in hours
Change of objective sleep measure (sleep onset latency, SOL) | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: sleep onset latency (SOL) in mins
Change in Objective Sleep Measures - Wake After Sleep Onset (WASO) | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: wake after sleep onset (WASO) in mins
Change in Objective Sleep Measures - Sleep Efficiency (SE) | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: sleep efficiency (SE), which is calculated by total sleep time divided by total time in bed, %
Change of Depressive Symptoms (Assessor-rated) | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Children's Depression Rating Scale (CDRS-R) is a 17-item rating scale based on a semistructured interview with children. Possible scores range from 17 to 113, with higher scores indicating severer depressive symptoms.
Change of Self-report states of depression and anxiety symptoms | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Hospital Anxiety and Depression Scale (HADS) is a self-assessed scale for detecting states of depression and anxiety. The depression subscale range in scores from 0 to 21, with higher scores indicating severer states of depression. Similarly, the anxiety subscale range in scores from 0-21 with higher scores indicating severer states of anxiety. No additional computation will be made with the two subscores.
Change of Self-report emotional states of depression, anxiety and stress | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Depression Anxiety Stress Scales consists of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS scales contains 14 items. Higher scores suggest more depression, anxiety and stress, respectively.
Change of Self-report depressive symptoms | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Beck's Depression Inventory (BDI) consists of 13 self-report items designed to measure depressive symptoms. Higher scores suggest high level of depression
Change of subjective mental well-being | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  The World Health Organisation- Five Well-Being Index (WHO-5) consists of 5 self-report items designed to measure subjective well-being. Higher scores indicate better well-being.
Change of dysfunctional beliefs and attitudes about sleep | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Dysfunctional Beliefs and Attitudes about Sleep (DBAS) is a 16-item self-rated scale measuring the respondent's sleep-related beliefs, more specifically, their expectations and attitudes regarding the causes, consequences, and potential treatments of sleep issues. A total score is calculated by averaging score of all items, possibly scored 0 to 10, with a higher score indicating more dysfunctional beliefs and attitudes about sleep.
Change of sleep hygiene and practice | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Sleep Hygiene Practice Scale (SHPS) is a 30-item self-rated scale measuring sleep hygiene behaviors, ranging in total scores from 30 to 180, with higher scores indicating lower levels of sleep hygiene.
Change of pre-sleep arousal | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Pre-Sleep Arousal Scale is a 16-item self-rated scale measuring pre-sleep arousal. There are two subscales on the cognitive and somatic manifestations of arousal, with eight items in each subscale (possibly scored from 8 to 40). In both cases, a higher score indicates higher pre-sleep arousal.
Change of sleep reactivity | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Ford Insomnia Response to Stress Test (FIRST) consists of 9 items designed to measure sleep reactivity. Possible scores range from 9 to 36. A higher score indicates higher sleep activity.
Change of Suicidal Ideation | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Depressive Symptom Inventory Suicidality Subscale (DSI-SS) is a 4-item self-rated scale measuring suicidal ideation. Possible total scores range from 0 to 12, with higher scores indicating higher suicidal ideation.
Change of Daytime Sleepiness | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Paediatric Daytime Sleepiness Scale (PDSS) is an 8-item self-rated scale measuring daytime sleepiness, ranging in total scores from 0 to 32 with higher scores indicating more sleepiness.
Change of Daytime Fatigue | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Multidimensional Fatigue Inventory (MFI) is a 20-item self-rated scale on fatigue symptoms. There are three subscales, measuring the physical (possibly scored from 7 to 35), mental (possibly scored from 6 to 30), and spiritual (possibly scored from 7 to 35), dimensions of fatigue. A grand total score can be calculated by summing up the three sub scores. In all cases, a higher score represents higher fatigue symptoms.
Change of Quality of Life (KIDSCREEN-27) | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  KIDSCREEN-27 is a 27-item self-rated scale measuring health related quality of life measure for children and adolescents. There are five subscales on: physical well-being (possibly scored from 5 to 25), psychological well-being (possibly scored 7 to 35), autonomy & parents (possibly scored 7 to 35), peers & social support (possibly scored 4 to 20), and school environment (possibly scored 4 to 20). A grand total score can be calculated by summing up the five sub scores. In all cases, a higher score represents higher perceived well-being.
Change of Overall Severity of Clinical Symptoms | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Clinical Global Impression (CGI) Scale is a clinician-rated scale, comprised of two one-item subscales: Severity of Illness (CGI-S) subscale evaluating the severity of psychopathology, and Clinical Global Improvement Scale (CGI-I) evaluating change from the initiation of treatment. In both cases, the score is given on a seven-point scale, with higher values indicating higher severity of illness and larger improvement respectively.
Change of Objective Cognitive Performance (visual attention & task switching) | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Trail Making Test for assessing visual attention and task switching. In Trail Making Test, longer reaction time indicates lower level of attention.
Change of Objective Cognitive Performance (inhibitory ability) | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Go/No-go Task for assessing inhibitory ability. In Go/No-go Task, a higher error rate indicates lower inhibition control.
Change of Objective Cognitive Performance (working memory by digit span) | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Digit Span Task for assessing working memory capacity. In Digit Span Task, a higher number of recalled digits indicates better working memory.
Change of Objective Cognitive Performance (working memory by N-Back) | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  N-back Task for assessing working memory capacity and manipulation. In N-back Task, a d prime score will be calculated based on the signal detection theory, where a higher score indicates better working memory performance.
Change of Objective Cognitive Performance (episodic memory) | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Chinese Auditory Verbal Learning Task for assessing episodic memory, where a higher number of recalled words indicates better episodic memory performance.
Change of Objective Cognitive Performance (problem solving) | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Wisconsin Card Sorting Test for assessing problem solving. In Wisconsin Card Sorting Test, lower executive functioning is indicated by a higher percentage of persistent errors and a higher number of trials taken to complete the first category.
Change of sleep related attention bias | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Sleep-related Dot-Probe Task for assessing sleep-related attention bias. In the Sleep-related Dot-probe Task, a higher attention bias score indicates higher vigilance towards sleep-related stimuli.
Change of risk-taking & decision making | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Balloon Analogue Risk Task for assessing risk-taking and decisionmaking. In Balloon Analogue Risk Task, a score will be calculated by averaging the number of pumps on unexploded blue balloons, where a higher score indicates more risk-taking and impulsive propensities.
Change of implicit cognition of suicide or death | Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants, and additional two follow-ups at Post-Treatment 6-month and Post-Treatment 12-month for participants in the treatment groups
  Suicide Implicit Association Test (IAT) for assessing implicit cognition of suicide or death. In the Suicide Implicit Association Test, positive D-scores indicate stronger implicit identification with death and negative D scores indicate stronger implicit identification with life
Change of emotion regulation abilities | Time Frame: Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants
  Difficulties in Emotion Regulation Scale (DERS) is a 36-item self-reported scale measuring emotion regulation problems. Every item uses a 1-to-5 Likert scale, with 1 represents "Almost never" and 5 represents "Almost always". Total score ranges from 36 to 180. Higher score represents higher difficulties in regulating emotions. Sub-scores will also be calculated on the following subscales:
  i. Nonacceptance of emotional responses ii. Difficulty engaging in goal-directed behavior iii. Impulse control difficulties iv. Lack of emotional awareness v. Limited access to emotion regulation strategies vi. Lack of emotional clarity
Change of emotion regulation tendency/capacity | Time Frame: Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants
  Emotion regulation questionnaire - frequency/capacity (ERQ-f/ERQ-c) is a 28-item scale designed to measure respondents' tendency/capacity to regulate their emotions in three ways: (1) Cognitive Reappraisal, (2) Expressive Suppression and (3) Distraction. Scores will be calculated separately for each subscale, ranging from 4 to 42. Each item will be answered on a 7-point Likert-type scale ranging from 1(strongly disagree) to 7 (strongly agree). For ERQ-f, higher score represents higher frequency of using certain regulation method. For ERQ-c, higher score represents higher capacity of using certain regulation method.
Change of ability/efficiency in using different emotion regulation strategies | Time Frame: Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants
  Emotion regulation task is a paradigm used to examined subjects' ability/efficiency in using different emotion regulation strategies (i.e., watch, reappraisal and distraction). Subject will first see a negative or neutral picture, followed by instructions on using which strategy to regulate their emotions induced by the picture (watch, reappraisal or distraction). There are four conditions: neutral-watch, negative-watch, negative-reappraisal, negative-distraction. After each picture, subjective emotional valence and arousal ratings (ranging from 1-9) will be collected. To examine the subjects' different emotion regulation ability, valence and arousal ratings will be analysed by comparing different conditions, groups, and time (pre/post-treatment).
Change of verbal fluency | Time Frame: Baseline, Post-Treatment (one-week after completion of the intervention/waiting period) for all participants
  Category Fluency Task will be used to assess verbal fluency. The total number of words produced will be summed and transformed into z-scores in comparison to local norms

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Xin Li, PhD,DClinPsy, Principal Investigator — The University of Hong Kong
Locations (1):
- Sleep Research Clinic and Laboratory, Department of Psychology, The University of Hong Kong, Hong Kong, Hong Kong